CLINICAL TRIAL: NCT05838196
Title: Does the Use of Point of Care Ultrasound During Inflammatory Bowel Disease Clinic Appointments Change Management, Speed up Treatment Decisions and Save Money: a Feasibility and Service Development Study
Brief Title: Service Development of POCUS in the IBD Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 155436
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Intestinal ultrasound
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participant will follow standard of care
- Point-of-care Ultrasound (Experimental): Participant will receive point-of-care ultrasound at time of clinic appointment and clinician will use result to inform treatment decision
  Interventions: Diagnostic Test: Point-of-care ultrasound

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound — Point-of-care ultrasound performed during clinic appointment
  Arms: Point-of-care Ultrasound

SUMMARY:
Study to determine whether the use of an ultrasound completed during an inflammatory bowel disease (IBD) clinic will speed up diagnosis, treatment initiation, reduce complications, save money and reduce investigations compared with our current standard of care.

DETAILED DESCRIPTION:
After being provided with study information and providing written informed consent, participants attending the inflammatory bowel disease clinic will be randomised to standard of care or to receiving an ultrasound during the clinic appointment. This ultrasound result will be used to determine treatment decisions. Participants will have a 6 month follow-up to capture outcome data and further medical record review will be conducted at one year.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or above
* Attending IBD clinic face-to-face
* Able to give informed consent.
* Belonging to one of the following groups:

  1. New patients with high clinical suspicion of IBD
  2. Known UC/IBD-U and possible flare
  3. Known Crohn's and possible flare
  4. Known IBD and assessing response to a new medication or following surgery
  5. Known IBD and clinician planning endoscopic or radiological investigations

Exclusion Criteria:

* Inflammatory bowel disease limited to proctitis with no clinical suspicion of extension

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Compare time to definitive IBD-related treatment initiation with the use of POCUS compared to standard of care | 6 months
  Time in days for when a new medication is started, dose changed, medication stopped, or surgery performed following the clinic appointment

SECONDARY OUTCOMES:
Does point of care ultrasound change clinical decision making in the IBD clinic | Immediate
  Does the clinical decision made before ultrasound differ from that following ultrasound.
Compare sensitivity and specificity of POCUS to identify active disease with standard of care investigations (MRI, ultrasound, endoscopy) | 6 months
  Using formalised imaging or endoscopy as gold standard for determining disease activity, compare findings on POCUS to determine sensitivity and specificity
Compare healthcare resource utilisation including outpatient appointments, need for further investigations and admissions in patients receiving POCUS or standard of care | 1 year
  Using NHS cost tariffs, estimated costs for participants following standard of care to those receiving POCUS over the year following enrolment
Compare findings at POCUS when performed by a gastroenterologist or a radiologist | 6 months
  POCUS will be performed by gastroenterologists or radiologist and outcomes on sensitivity/specificity will be compared between the two
Compare clinical disease activity scores when POCUS is used compared with standard of care | 6 months
  Using disease activity score questionnaires (HBI (If Crohn's disease) or SCCAI (If ulcerative Colitis)) at baseline and six months.
Compare use of steroids with POCUS compared with standard of care | 1 year
  Number of courses of steroids and total steroid dose over the duration of the trial
Compare haemaglobin levels when POCUS is used compared with standard of care | 6 months
  Are there significant difference between the change in haemaglobin from baseline to six months in the POCUS group compared with standard of care
Compare CRP levels when POCUS is used compared with standard of care | 6 months
  Are there significant difference between the change in CRP from baseline to six months in the POCUS group compared with standard of care
Compare Platelets when POCUS is used compared with standard of care | 6 months
  Are there significant difference between the change in platelets from baseline to six months in the POCUS group compared with standard of care

CONTACTS AND LOCATIONS:
Overall Officials: William Blad, BM BCh, Principal Investigator — University College London Hospitals Trust
Locations (1):
- University College London Hospitals NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No